CLINICAL TRIAL: NCT04801992
Title: Retrospective, Observational, Monocenter And Single-Arm Trial Following Subjects Bilaterally Implanted With Mini Well Ready For 2 Years After The Second Eye Implant
Brief Title: Trial Following Subjects Bilaterally Implanted With Mini Well Ready For 2 Years After the Second Eye Implant
Status: Completed | Type: Observational
Sponsor: SIFI SpA (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Other Study IDs: PSM8 Sub-study
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Cataract
Keywords: Cataract surgery; Extended Depth-of-Focus (EDOF); Intraocular Lens (IOL); Presbyiopa correction
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MINI WELL Ready (SIFI SpA, Italy): Extended depth of focus intraocular lens implantation
  Interventions: Device: MINI WELL Ready (SIFI SpA, Italy)

INTERVENTIONS:
Device: MINI WELL Ready (SIFI SpA, Italy) — Implantation during cataract surgery of the progressive extended depth of focus intraocular lens for the posterior chamber to replace the crystalline lens in the correction of aphakia in adult patients.

SUMMARY:
The study objective is to evaluate the visual performance of MINI WELL Ready at 24 months following the second eye implant. The objectives of safety are to evaluate the rate of Secondary Surgical Interventions related to the optical properties of the IOL for first and second operative eye separately at 24 months and the rate of visual disturbances and distortions as reported by the subjects as detected by using the Halo & Glare Simulator.

DETAILED DESCRIPTION:
The present post-.market follow-up study (PSM8 sub-study) is an ancillary study of the PSM8 post market clinical trial (NCT02740010)

ELIGIBILITY:
Inclusion Criteria:

• Previous enrolment in the PSM8 study in the period from March, 1st 2014 to March, 31st 2016 with the following:

* Any gender and age above 18 years.
* Cataract or Refractive Lens Exchange (RLE) surgery; will be included patients submitted to conventional phacoemulsification as to femtolaser procedure; no specification regarding corneal incision size and position.
* Symmetrical preoperative keratometric astigmatism < 1.00 D.
* Healthy corneas, not surgically treated

Exclusion Criteria:

* Previous corneal surgery (i.e. pterygium, refractive surgery).
* Eye diseases with visual acuity < 20/32.
* Pseudoexfoliation.
* Abnormal pupil size and position.
* Use of contact lens 30 days before the preoperative visit.
* Corneal warpage.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects affected by cataract that fulfill eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Subjective Refraction | 26 months
Binocular Defocus Curve | 26 months
  Binocular Defocus Curve (+2.0 D to -4.0 D in 0.5 D increments)
UDVA | 26 months
  Monocular and Binocular Uncorrected Distance Visual Acuity (UDVA) at 4m
CDVA | 26 months
  Monocular and Binocular Corrected Distance Visual Acuity (CDVA) at 4m
UIVA at 100 cm | 26 months
  Monocular and Binocular Uncorrected Intermediate Visual Acuity at 100 cm (100% and 10% contrast)
DCIVA at 100 cm | 26 months
  Monocular and Binocular Distance Corrected Intermediate Visual at 100 cm (100% and 10% contrast)
UIVA at 60 cm | 26 months
  Monocular and Binocular Uncorrected Intermediate Visual Acuity at 60 cm (100% and 10% contrast)
DCIVA at 60 cm | 26 months
  Monocular and Binocular Distance Corrected Intermediate Visual Acuity at 60 cm (100% and 10% contrast)
UNVA | 26 months
  Monocular and Binocular Uncorrected Near Visual Acuity at 40cm (100% contrast)
DCNVA | 26 months
  Monocular and Binocular Distance Corrected Near Visual Acuity at 40cm (100% contrast)
Contrast Sensitivity | 26 months
  Binocular Contrast Sensitivity with correction for distance
Reading Performance | 26 months
  Binocular Reading Performance with and without correction for distance
VR-11R | 26 months
  Visual Function -11R Questionnaire from 4 (without difficulties) to 0 (performance impossible due to difficulties)

SECONDARY OUTCOMES:
Postoperative Complications Rate of postoperative complication | 26 months
Subjective Posterior Capsule Opacification | 20-26 months
  Subjective assessment through slit lamp
Posterior Capsulotomy | 26 months
Adverse Events including SSIs | 26 months
Device Deficiencies | 26 months
  Descriptive assessment
Photic Phenomena Assessment | 26 months
  Using the Halo and Glare Simulator software

CONTACTS AND LOCATIONS:
Locations (1):
- U.O. Oftalmologia I Dipartimento di Scienze Mediche di Base, Neuroscienze e Organi di Senso Università degli Studi di Bari "Aldo Moro", Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jiang T, Jiang J, Zhou Y, Zhao GQ, Li H, Zhao SY. Cataract surgery in aged patients: phacoemulsification or small-incision extracapsular cataract surgery. Int J Ophthalmol. 2011;4(5):513-8. doi: 10.3980/j.issn.2222-3959.2011.05.11. Epub 2011 Oct 18. PMID 22553713
- [Result] Packer M, Fine IH, Hoffman RS. Aspheric intraocular lens selection: the evolution of refractive cataract surgery. Curr Opin Ophthalmol. 2008 Jan;19(1):1-4. doi: 10.1097/ICU.0b013e3282f2d791. No abstract available. PMID 18090888
- [Result] Kohnen T, Klaproth OK, Buhren J. Effect of intraocular lens asphericity on quality of vision after cataract removal: an intraindividual comparison. Ophthalmology. 2009 Sep;116(9):1697-706. doi: 10.1016/j.ophtha.2009.03.052. Epub 2009 Jul 29. PMID 19643497
- [Result] Becker KA, Martin M, Rabsilber TM, Entz BB, Reuland AJ, Auffarth GU. Prospective, non-randomised, long term clinical evaluation of a foldable hydrophilic single piece intraocular lens: results of the Centerflex FDA study. Br J Ophthalmol. 2006 Aug;90(8):971-4. doi: 10.1136/bjo.2006.092437. Epub 2006 May 10. PMID 16687454
- [Result] Lehmann R, Waycaster C, Hileman K. A comparison of patient-reported outcomes from an apodized diffractive intraocular lens and a conventional monofocal intraocular lens. Curr Med Res Opin. 2006 Dec;22(12):2591-602. doi: 10.1185/030079906X158039. PMID 17166341
- [Result] Leyland M, Zinicola E. Multifocal versus monofocal intraocular lenses in cataract surgery: a systematic review. Ophthalmology. 2003 Sep;110(9):1789-98. doi: 10.1016/S0161-6420(03)00722-X. PMID 13129879
- [Result] Steinert RF. Visual outcomes with multifocal intraocular lenses. Curr Opin Ophthalmol. 2000 Feb;11(1):12-21. doi: 10.1097/00055735-200002000-00004. PMID 10724823
- [Result] Blaylock JF, Si Z, Vickers C. Visual and refractive status at different focal distances after implantation of the ReSTOR multifocal intraocular lens. J Cataract Refract Surg. 2006 Sep;32(9):1464-73. doi: 10.1016/j.jcrs.2006.04.011. PMID 16931257